CLINICAL TRIAL: NCT01147653
Title: Is Autologous Umbilical Cord Blood Reinfusion Beneficial in Children With Cerebral Palsy: A Randomized, Blinded, Placebo-Controlled, Crossover Study
Brief Title: A Randomized Study of Autologous Umbilical Cord Blood Reinfusion in Children With Cerebral Palsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Joanne Kurtzberg, MD (Other)
Collaborators: The Robertson Foundation (Other)
Responsible Party: Sponsor-Investigator, Joanne Kurtzberg, MD, Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00017801
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Results first posted 2017-06-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy; CP; Spastic Cerebral Palsy
Keywords: Cerebral Palsy; CP; Spastic Cerebral Palsy; Cord Blood; Umbilical Cord Blood; Autologous Cord Blood
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous UCB Reinfusion First,Then Placebo (Active Comparator): Subjects receive their autologous umbilical cord blood cells at Baseline, than placebo at Year 1.
  Interventions: Biological: Autologous UCB Reinfusion; Other: Placebo
- Placebo First, Then Autologous UCB Reinfusion (Placebo Comparator): Subjects receive placebo at Baseline, then autologous umbilical cord blood cell reinfusion at Year 1.
  Interventions: Biological: Autologous UCB Reinfusion; Other: Placebo

INTERVENTIONS:
Biological: Autologous UCB Reinfusion — Autologous umbilical cord blood (UCB) reinfusion
Other: Placebo — Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of a single intravenous infusion of autologous umbilical cord blood (UCB) for the treatment of pediatric patients with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy results from in utero or perinatal injury to the developing brain, often through stroke, hypoxic insult or hemorrhage. Currently available treatments for patients with cerebral palsy are supportive, but not curative. Umbilical cord blood (UCB) has been shown to lessen the clinical and radiographic impact of hypoxic brain injury and stroke in animal models. UCB also engrafts and differentiates in brain, facilitating neural cell repair, in animal models and human patients with inborn errors of metabolism undergoing allogeneic, unrelated donor UCB transplantation. We hypothesize that, in the setting of brain injury, infusion of autologous UCB will facilitate neural cell repair resulting in improved function in pediatric patients with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months and ≤ 6 years
* Diagnosis: Spastic cerebral palsy with diplegia, hemiplegia, or quadraplegia.
* Performance status:

Gross Motor Function (GMF) Classification Score levels II - IV or GMF Score leve I, age >/= 2 years Spastic hemiplegia: GMF Score II-IV or minimal functional capabilities in the affected upper extremity. A subject classified as GMFCS level I with significant upper extremity impairment will be eligible if the affected upper extremity is used as an assist only. An eligibility committee will meet to review the child's records and determine eligibility.

Bilateral hypotonic CP (diplegia or quadriplegia): GMF Score II-IV and an abnormal brain MRI suggestive of an acquired etiology (versus a genetic etiology or brain malformation).

* Autologous umbilical cord blood available at a private or public cord blood bank with a minimum total nucleated cell dose of ≥ 1 x 107 cells/kilogram.
* Parental consent.

Exclusion Criteria:

* Athetoid cerebral palsy.
* Autism and autistic spectrum disorders without motor disability.
* Hypsarrhythmia.
* Intractable seizures causing epileptic encephalopathy.
* Evidence of a progressive neurologic disease.
* Known HIV or uncontrolled bacterial, fungal, or viral infections.
* Impaired renal or liver function as determined by serum creatinine >1.5mg/dL and/or total bilirubin >1.3mg/dL.
* Head circumference >3 standard deviations below the mean for age.
* Known genetic disease or phenotypic evidence of a genetic disease on physical examination.
* Concurrent genetic or acquired disease or comorbidity(ies) that could require a future allogeneic stem cell transplant.
* Requires ventilatory support, including home ventilator, CPAP, BiPAP, or supplemental oxygen.
* Patient's medical condition does not permit safe travel.
* Previously received any form of cellular therapy.
* Autologous umbilical cord blood unit has any of the following:

  1. Total nuclear cell dose < 1 x 107 cells/kilogram
  2. Positive maternal infectious disease markers (except CMV)
  3. Evidence of infectious contamination of the cord blood unit
  4. Lack of a test sample to confirm identity
  5. Evidence of a genetic disease
* Unable to obtain parental consent.

Ages: 12 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2010-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Kurtzberg, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Sun JM, Song AW, Case LE, Mikati MA, Gustafson KE, Simmons R, Goldstein R, Petry J, McLaughlin C, Waters-Pick B, Chen LW, Wease S, Blackwell B, Worley G, Troy J, Kurtzberg J. Effect of Autologous Cord Blood Infusion on Motor Function and Brain Connectivity in Young Children with Cerebral Palsy: A Randomized, Placebo-Controlled Trial. Stem Cells Transl Med. 2017 Dec;6(12):2071-2078. doi: 10.1002/sctm.17-0102. Epub 2017 Oct 28. PMID 29080265

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled and randomized on the same day.
Groups:
- Autologous UCB Reinfusion First, Then Placebo: Subjects receive autologous umbilical cord blood at Baseline, then Placebo at Year 1.
- Placebo First, Then Autologous UCB Reinfusion: Subjects receive Placebo at Baseline, then autologous umbilical cord blood at Year 1.
Period: Year 1
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Started | 32 | 31
Completed | 32 | 31
Not Completed | 0 | 0
Period: Year 2
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Started | 32 | 31
Completed | 30 | 28
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Autologous UCB First, Then Placebo: Subjects receive autologous umbilical cord blood at Baseline, then Placebo at Year 1.
- Total: Total of all reporting groups
Arm/Group | Autologous UCB First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Median (Full Range); unit: Years] | 2.1 [1.1 to 6.2] | 2.3 [1.1 to 7.0] | 2.3 [1.1 to 7.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 20 | 22 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 27 | 28 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
GMFCS Level [Count of Participants; unit: Participants] — The Gross Motor Function Classification System (GMFCS) classifies gross motor function of children with cerebral palsy into Levels I (least disabled) to V (most disabled). For example, children at Level I are able to walk at home, in school, and in the community and can climb stairs without a railing. At Level II children may walk with assistance and can climb stairs using a railing. At Level III children walk with handheld assistive devices for short distances but use a wheelchair for long distance mobility. Mobility at Levels IV and V require physical assistance or powered devices.
  Participants
    Level I | 11 | 6 | 17
    Level II | 9 | 15 | 24
    Level III | 4 | 4 | 8
    Level IV | 8 | 6 | 14
Type of Cerebral Palsy [Count of Participants; unit: Participants]
  Spastic Diplegia | 6 | 6 | 12
  Spastic Hemiplegia | 15 | 15 | 30
  Spastic Quadriplegia | 10 | 7 | 17
  Hypotonic Quadriplegia | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Gross Motor Function Measure 66 (GMFM-66) Score
Description: Change in Gross Motor Function Measure 66 (GMFM-66) Score from Baseline to Year 1. The GMFM-66 is a clinical tool used to evaluate gross motor function in children with cerebral palsy and is scored using a propriety software program called the Gross Motor Ability Estimator (GMAE) that produces an interval level continuous score ranging from 0 to 100. Higher scores indicate better motor function. A negative change in GMFM-66 score indicates a reduction in motor function, a positive change indicates improvement in motor function, and zero indicates no change in motor function.
Time Frame: Baseline to Year 1
Population: All enrolled patients were analyzed as randomized from Baseline to Year 1.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Autologous UCB Reinfusion First, Then Placebo: Subjects receive their autologous umbilical cord blood cells at Baseline, than placebo at Year 1.
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 32 | 31
units on a scale | 7.5 (6.8) | 6.9 (5.6)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The true mean 1-year change in GMFM-66 is the same on Autologous Umbilical Cord Blood and Placebo; Test type: Superiority; p = 0.72, t-test, 2 sided; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.6 to 3.7]

2. Secondary Outcome: Change in Peabody Gross Motor Quotient From Baseline to Year 1
Description: The Peabody Developmental Motor Scales - Second Edition (PDMS-2) measures gross and fine motor skills in children from birth through five years of age. The Gross Motor Quotient score from the PDMS-2 was used in this study to evaluate gross motor function. The Gross Motor Quotient measures the ability to use large muscle systems for locomotion, maintain a stable posture when not moving, and throw/catch objects. The range of possible scores is 41 to 164. High scores indicate better gross motor function. Lower scores indicate less gross motor function ability. The change in Gross Motor Quotient from Baseline to Year 1 was evaluated in this study. Positive numbers indicate an increase in gross motor ability, negative numbers indicate decreases in gross motor function, and a zero indicates no change.
Time Frame: Baseline to Year 1
Population: Participants outside of the applicable age range for the PDMS-2 at Baseline or Year 1 were excluded from the analysis.
Measure: Median (Full Range); unit: units on a scale
Groups:
- Autologous Umbilical Cord Blood Reinfusion: Subjects receive their autologous umbilical cord blood cells at Baseline, than placebo at Year 1.
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 24 | 26
units on a scale | 1 [-10 to 20] | -0.5 [-19 to 15]
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Change in IT-QOL Questionnaire Score
Description: The Infant and Toddler Quality of Life Questionnaire (IT-QOL) was utilized for children ages one to three years at study entry.This 97-item questionnaire is completed by the parents and covers 12 concepts related to the physical, mental, and social well being of the child and the impact of their illness on the family. Scores range from 0 (worst health) to 100 (best health). The change from Baseline to Year 1 is summarized here for each of the 12 items on the questionnaire. Negative values indicate a decline in quality of life over time, positive values indicate an improvement, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: The analysis includes patients whose parents reported scores on each item at both Baseline and Year 1 and whose children met the age criteria for the questionnaire at both time points.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 24 | 21
units on a scale
  Behavior | 4.5 [-13 to 20] | 3 [-15 to 20]
  Bodily Pain/Discomfort | 0 [-42 to 42] | 8 [-25 to 25]
  Family Cohesion | 0 [-40 to 40] | 0 [-25 to 25]
  General Behavior | 4 [-35 to 29] | 2 [-21 to 28]
  General Health Perceptions | 0 [-23 to 21] | 0 [-19 to 25]
  Global Behavior | 0 [-40 to 55] | 0 [-55 to 30]
  Growth and Development | 7.5 [-22 to 35] | 3 [-28 to 30]
  Overall Health | 0 [-30 to 30] | 0 [-40 to 25]
  Parental Impact-Emotional | 18 [-14 to 50] | 0 [-21 to 53]
  Parental Impact-Time | 2 [-22 to 43] | 0 [-43 to 47]
  Physical Abilities | 5.50 [-15 to 35] | 6 [-33 to 34]
  Temperament and Moods | 4 [-20 to 25] | 2 [-8 to 30]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Behavior change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.473, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Bodily Pain/Discomfort change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.377, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Family Cohesion change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.844, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month General Behavior change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.322, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month General Health Perceptions change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.927, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Global Behavior change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.199, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Growth and Development change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.294, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Overall Health change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.726, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Parental Impact-Emotional change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.315, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Parental Impact-Time change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.396, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Physical Abilities change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.381, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Temperament and Moods change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.869, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in CP-QOL Score
Description: Children age four years or older at study entry were assessed using the disease-specific "CP-QOL Child" assessment tool as completed by a parent. The CP-QOL Child primary-caregiver proxy form is designed for children 4 - 12 with cerebral palsy and contains 66 items which assess physical, emotional, and social well being as well as access to services and acceptance by others. Scores are summarized in seven topic areas. Scores in each area range from 0 (worst health) to 100 (best health). The change score from Baseline to Year 1 is summarized here for each item. Negative scores indicated a decrease in quality of life, positive scores indicate an increase and zero indicates no change.
Time Frame: Baseline, Year 1
Population: as for outcome 3
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 6 | 5
units on a scale
  Access to services | -13 [-32 to 12] | 15 [-13 to 28]
  Emotional well being and self esteem | -8.5 [-30 to 4] | 10 [-13 to 90]
  Family Health | -3.5 [-37 to 3] | 0 [-18 to 19]
  Functioning | -11.5 [-22 to 6] | 3 [-14 to 30]
  Pain and impact of disability | 7 [-17 to 17] | -5 [-22 to 3]
  Participation and physical health | -3 [-20 to 12] | 17 [-20 to 35]
  Social wellbeing and acceptance | -4 [-11 to 4] | 3 [-17 to 12]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12 month Access to Services change score is identically distributed in patients assigned Autologous Cord Blood Reinfusion First and Placebo First; Test type: Superiority; p = 0.055, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month 2 Emotional Well Being and Self Esteem change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.121, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month 2 Family Health change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.647, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Functioning change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.170, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Pain and Impact of Disability change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.410, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Participation and Physical Health change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.200, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The 12-month Social wellbeing and acceptance change score is identically distributed in patients assigned Autologous UCB Reinfusion First and Placebo First; Test type: Superiority; p = 0.225, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Whole Brain Connectivity Measured by Diffusion Tensor Magnetic Resonance Imaging (MRI)
Description: Change in number of connections in the brain as measured by diffusion tensor magnetic resonance imaging (MRI). Changes in connectivity are normalized to white matter volume of the brain. A positive number indicates an increase in connections, a negative number indicates a decrease, and zero indicates no change. The number of connections is expressed in terms of 10e5. For example, a change of 1 indicates an increase of 1x10e5 or 100,000 connections.
Time Frame: Baseline to Year 1
Population: Patients without substantial morphologic brain abnormalities that prevented accurate anatomical image parcellation.
Measure: Median (Full Range); unit: Number of connections x10e5
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 23 | 15
Number of connections x10e5 | 0.3 [-0.5 to 0.6] | 0.2 [-0.5 to 0.6]

6. Secondary Outcome: Change in Loes Score of Functional MRI From Baseline to Year 1 and From Year 1 to Year 2
Description: No data were collected from this procedure because enrolled subjects who were eligible to receive fMRI were unable to comply with the procedure.
Time Frame: Baseline, Year 1, Year 2
Population: No data was available.
Groups:
- Autologous UCB Reinfusion First,Then Placebo: Subjects receive their autologous umbilical cord blood cells first, than placebo at Year 1.
- Placebo First, Then Autologous UCB Reinfusion: Subjects receive placebo first, then autologous umbilical cord blood cell reinfusion at Year 1.
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Bayley Scales of Infant and Toddler Development-III, Cognitive Composite From Baseline to Year 1
Description: Cognitive function was assessed in English-speaking study participants using one of three different tools depending on the age of the patient at the time of assessment: The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), the Wechsler Intelligence Scale for Children (WISC-IV), and the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III). Some patients were assessed with different tools at subsequent visits as they aged during the conduct of the trial. The Bayley-III is designed to assess developmental functioning of infants and toddlers. Scores for the Cognitive Composite range from 1 to 19 and results in the range of 8 to 12 are considered average. The outcome measure reported here is the change in Cognitive Composite between Baseline to Year 1. Positive numbers indicate increases in cognitive functioning, negative numbers indicate a decrease, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: The Bayley III is an age-specific test and was used for 42 patients at Baseline. A total of 27 of these patients were also scored with the Bayley III at Year 1. The results here represent change from Baseline to Year 1 in the 27 participants assessed with the Bayley III at both time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 14 | 13
units on a scale | 3.2 (3.0) | 8.1 (3.3)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.290, t-test, 2 sided

8. Secondary Outcome: Change in Wechsler Preschool and Primary Scale of Intelligence (WPPSI) III Full Scale Intelligence Quotient (IQ) for Younger Children (Ages 2 Years & 6 Months to 3 Years & 11 Months) From Baseline to Year 1.
Description: Cognitive function was assessed in English-speaking study participants using one of three different tools depending on the age of the patient at the time of assessment: The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), the Wechsler Intelligence Scale for Children (WISC-IV), and the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III). Some patients were assessed with different tools at subsequent visits as they aged during the conduct of the trial. There are two versions of the WPPSI-III for two different age ranges: 2 years & 6 months to 3 years & 11 months, and 4 years to 7 years & 3 months. The Full Scale IQ is calculated for both age ranges and provides a continuous score with an average of 100 and a standard deviation of 15. Change from Baseline to Year 1 was evaluated, with positive numbers indicating an increase in cognitive ability, negative numbers indicating a decrease in cognitive ability, and zero indicating no change.
Time Frame: Baseline to Year 1
Population: Change scores were evaluable in only 2 subjects who were assessed with the WPPSI-III at both Baseline and Year 1. One subject was randomized to Autologous Cord Blood and the other to Placebo.
Measure: Number; unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 1 | 1
units on a scale | 14 | -8

9. Secondary Outcome: Change in the Wechsler Intelligence Scale for Children (WISC-IV) From Baseline to Year 1.
Description: Cognitive function was assessed in English-speaking study participants using one of three different tools depending on the age of the patient at the time of assessment: The Bayley Scales of Infant and Toddler Development, Third Edition (Bayley-III), the Wechsler Intelligence Scale for Children (WISC-IV), and the Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III). Some patients were assessed with different tools at subsequent visits as they aged during the conduct of the trial. The WISC-IV is designed for children 6 years 0 months to 16 years 11 months. This study used the Full Scale IQ, which ranges from 45 to 155 with a mean of 100 and standard deviation of 15. Higher scores indicate stronger cognitive function. Scores between 90 and 110 are considered to be within the range of average IQ.
Time Frame: Baseline to Year 1
Population: Only one patient in this trial was evaluated with the WISC-IV and thus change over time could not be evaluated using this outcome measure. The single value for this patient is reported here.
Measure: Number; unit: Full Scale IQ Points
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 0 | 1
Full Scale IQ Points |  | 103

10. Secondary Outcome: Change in Cognitive Z-Score From Baseline to Year 1
Description: Because patients in this study were evaluated with different cognitive assessments based on their age at the time of assessment (The Bayley-III Cognitive Composite, the WPSSI-III Full Scale IQ, and the WISC-IV Full Scale IQ Composite), with some patients being assessed using different tools at subsequent visits during the trial, a method for combining the assessments was employed to evaluate change in cognitive function over time in as many patients as possible. A cognitive Z-score was calculated for each participant at Baseline and Year 1 by adjusting each score by the relevant assessments' population mean and standard deviation. The Z-scores represent the distance from the population mean, as measured by standard deviations. The analysis presented here summarizes the change in Z-score between Baseline and Year 1. A positive number indicates an increase in cognitive function, a negative number indicates a decrease, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: When using all available cognitive assessments, the change in cognitive Z-score was available for 42 of the 63 participants.
Measure: Mean (Standard Error); unit: Z scores
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 21 | 21
Z scores | 0.2 (0.2) | 0.3 (0.2)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.697, t-test, 2 sided

11. Secondary Outcome: Change in Assisting Hand Assessment (AHA) Score From Baseline to Year 1
Description: The Assisting Hand Assessment (AHA) measures the use of hemiplegic cerebral palsy patients' involved hand in tasks involving two hands. The test is valid for ages 18 months to 12 years. The score is an interval scale ranging from 22 to 88 with higher numbers indicating more effective use of the affected hand in performance of bimanual tasks. Change in this score was evaluate between Baseline and Year 1. Positive numbers indicate more effective use of the affected hand, negative numbers indicate a reduction in the effective use of the affected hand, and a zero indicates no change.
Time Frame: Baseline to Year 1
Population: Participants who were less than 18 months old, or had diplegia or quadriplegia were excluded. For those with unspecified typography, AHA scores were excluded if scores on either the Modified Ashworth Scale or Barry-Albright Dystonia scale indicated neither or both of the upper extremities were involved.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 9 | 10
units on a scale | 5.4 (2.1) | 5.1 (2.3)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.912, t-test, 2 sided

12. Secondary Outcome: Change in Pediatric Evaluation of Disability (PEDI) Self Care Score
Description: The Pediatric Evaluation of Disability is used to evaluate functional skills in children aged 6 months to 7 years in three areas: Self Care, Mobility, and Social Function. The score in each area can range from 10-90. Higher scores indicate higher function. The change from Baseline to Year 1 in the Self Care score is presented here. Positive scores indicate increased function, negative scores indicate a decrease, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: Patients were excluded if change scores were not observable due to missing data at Baseline or Year 1.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 31 | 29
units on a scale | -3.7 (2) | -2.2 (1.4)
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.544, t-test, 2 sided

13. Secondary Outcome: Change in Pediatric Evaluation of Disability (PEDI) Mobility Score
Description: The Pediatric Evaluation of Disability is used to evaluate functional skills in children aged 6 months to 7 years in three areas: Self Care, Mobility, and Social Function. The score in each area can range from 10-90. Higher scores indicate higher function. The change from Baseline to Year 1 in the Mobility score is presented here. Positive scores indicate increased function, negative scores indicate a decrease, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: Patients were excluded if change scores were not observable due to missing data at Baseline or Year 1.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 31 | 29
units on a scale | 0 [-21.81 to 19.80] | 0 [-18.50 to 13.21]
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Change in Pediatric Evaluation of Disability (PEDI) Social Function Score
Description: The Pediatric Evaluation of Disability is used to evaluate functional skills in children aged 6 months to 7 years in three areas: Self Care, Mobility, and Social Function. The score in each area can range from 10-90. Higher scores indicate higher function. The change from Baseline to Year 1 in the Social Function score is presented here. Positive scores indicate increased function, negative scores indicate a decrease, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: Patients were excluded if change scores were not observable due to missing data at Baseline or Year 1.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 31 | 29
units on a scale | -0.5 (2.0) | -1.3 (1.8)
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.76, t-test, 2 sided

15. Secondary Outcome: Change in Child Behavior Checklist (CBCL) Z-score Internalizing Problems From Baseline to Year 1
Description: Two versions of the CBCL exist for children ages 1.5 to 5 years and ages 6-18 years. The CBCL evaluates internalizing and externalizing behaviors and total problems using 99-item assessments that are scored on an ordinal scale as 0 for "not true of the child," 1 for "somewhat or sometimes true of the child," and 2 for "very true or often true of the child" based on behavior in the preceding two months. Scores are expressed on a standard normal distribution with mean 50 and standard deviation 10. Z scores were created for analysis. A Z-score represents the distance from the population mean in terms of the number of standard deviations. The change in Z-score from Baseline to Year 1 was calculated for each patient. A positive number indicates an increase in the behavior, a negative number indicates a decrease in the behavior, and a zero indicates no change.
Time Frame: Baseline to Year 1
Population: Evaluations done outside the age ranges specified for the assessments were excluded, the majority being assessments that were done on patients who were not yet 1.5 years of age.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 23 | 22
units on a scale | -0.6 [-1.8 to 2.5] | 0.0 [-2.2 to 1.0]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.176, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change in Child Behavior Checklist (CBCL) Z-score Externalizing Problems From Baseline to Year 1
Description: as for outcome 15
Time Frame: Baseline to Year 1
Population: as for outcome 15
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 23 | 22
units on a scale | -0.2 (0.2) | 0.1 (0.1)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.099, t-test, 2 sided

17. Secondary Outcome: Change in Child Behavior Checklist (CBCL) Z-score Total Problems From Baseline to Year 1
Description: as for outcome 15
Time Frame: Baseline to Year 1
Population: as for outcome 15
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 23 | 22
units on a scale | -0.3 [-2.0 to 2.8] | 0.1 [-1.9 to 1.2]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.131, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Change in Parental Distress From Baseline to Year 1
Description: Parent stress was evaluated with the Parenting Stress Index - Short Form for children aged 0-12 years, which measures stress in three domains: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. Results in each domain are expressed as percentiles. Scores from the 15th-80th percentile are considered to be within the normal range.
  Scores at or above the 85th percentile considered high distress. Scores greater than the 89th percentile indicate clinically significant levels of distress. Analysis focused on changes in percentile scores between Baseline and Year 1. Positive numbers represent an increase in distress, negative numbers represent a decrease in distress, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: No participants were outside the age range for this test but change scores could not be calculated for some participants due either to missing data at the Baseline or Year 1 visit.
Measure: Mean (Standard Error); unit: Change in percentile score
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 28 | 29
Change in percentile score | 1.0 (4.5) | -3.6 (4.6)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.478, t-test, 2 sided

19. Secondary Outcome: Change in Parent-Child Dysfunctional Interaction From Baseline to Year 1
Description: as for outcome 18
Time Frame: Baseline to Year 1
Population: as for outcome 18
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 28 | 29
units on a scale | 0.0 [-35.0 to 45.0] | -10.0 [-56.0 to 41.0]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.029, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change in Difficult Child Score From Baseline to Year 1
Description: as for outcome 18
Time Frame: Baseline to Year 1
Population: as for outcome 18
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 28 | 29
units on a scale | -0.2 (4.8) | 6.9 (5.0)
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.310, t-test, 2 sided

21. Secondary Outcome: Modified Ashworth Scale at Baseline
Description: The Modified Ashworth Scale uses a 6 point scale (range 0, 1, 1+, 2, 3, or 4) to measure spasticity in 5 body regions (central, right upper extremity, left upper extremity, right lower extremity, and left lower extremity). Scores of 0 indicate no increase in muscle tone whereas a score of 4 indicates rigidity in flexion or extension.
Time Frame: Baseline
Population: Patients are classified by their maximum score, regardless of body region.
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 30 | 30
Participants
  0 @ Baseline | 2 | 3
  1 @ Baseline | 4 | 3
  1+ @ Baseline | 5 | 3
  2 @ Baseline | 11 | 11
  3 @ Baseline | 8 | 8
  5 @ Baseline | 0 | 2

22. Secondary Outcome: Modified Ashworth Scale at Year 1
Description: as for outcome 21
Time Frame: Year 1
Population: Patients are classified by their maximum score, regardless of body region.
Measure: Count of Participants; unit: Participants
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 31 | 30
Participants
  0 @ Year 1 | 1 | 1
  1 @ Year 1 | 3 | 5
  1+ @ Year 1 | 6 | 8
  2 @ Year 1 | 10 | 9
  3 @ Year 1 | 10 | 6
  4 @ Year 1 | 1 | 1
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The population distribution of Modified Ashworth Scale scores is the same at 1-year post-infusion with autologous cord blood and placebo; Test type: Superiority; p = 0.233, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Change in Bruininks-Oseretsky-2 Total Motor Composite From Baseline to Year 1
Description: The Bruininks-Oseretsky Test of Motor Proficiency, Second Edition, (BOT-2) evaluates motor function in four areas: stability, mobility, strength, coordination, and object manipulation. A Total Motor Composite is then calculated and expressed on a normal distribution with mean 50 and standard deviation of 10. Higher scores indicate better motor function. The BOT-2 Total Motor Composite was used to measure motor function in children at age 6 in this study. The study intended to evaluate change in the BOT-2 Total Motor Composite from Baseline to Year 1, where positive change indicates improvement in motor function, negative change indicates decrease in motor function, and zero indicates no change.
Time Frame: Baseline to Year 1
Population: The BOT-2 Total Motor Composite was available at Baseline and Year 1 in only 1 subject. The change score for that subject is reported here.
Measure: Number; unit: units on a scale
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 1 | 0
units on a scale | -1 |

24. Secondary Outcome: Correlation Between Clinical Response and RNA Expression of Neural, Endothelial and Inflammatory Cytokines Measured by RNA Arrays in Cord Blood Cells Given to These Patients.
Description: Various pre-selected neural, angiogenic, and anti-inflammatory markers expressed by UCB cells and clinical response will be evaluated.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2028-06

25. Secondary Outcome: Parent Experience of Child Illness (PECI)
Description: The PECI is a 25-item measure designed to examine parental adjustment related to caring for a chronically ill child.
Time Frame: Baseline to Year 1
Population: Data not collected due to the measure not being validated for children with Cerebral Palsy.
Groups:
- Autologous UCB Reinfusion First, Then Placebo: Subjects receive their autologous umbilical cord blood cells at Baseline, then placebo at Year 1.
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 0 | 0

26. Other Pre Specified Outcome: Change in Barry-Albright Dystonia Total Score From Baseline to Year 1
Description: The Barry-Albright Dystonia Scale measures generalized dystonia in eight body regions (eyes, mouth, neck, trunk, and the four extremities) using an ordinal scale (0=no dystonia, 1=slight dystonia, 2=mild dystonia, 3=moderate dystonia, and 4=severe dystonia). Individual scores for each region are summed to obtain a total score. The total score can range from 0 to 32 and higher scores indicate an overall greater degree of dystonia. The change in Barry-Albright Dystonia Total Score was evaluated from Baseline to Year 1. Positive numbers indicate increasing dystonia, negative numbers indicate a decrease in dystonia, and zero indicates no change.
Time Frame: Baseline to Year 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First,Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 32 | 31
units on a scale | 0.0 [-12.0 to 10.0] | 0.0 [-11.0 to 28.0]
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First,Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; Test type: Superiority; p = 0.762, Wilcoxon (Mann-Whitney)

27. Post Hoc Outcome: Gross Motor Function Measure 66 (GMFM-66) Change Score at 1 Year by Infused Dose
Description: Gross Motor Function Measure 66 (GMFM-66) Change Score at 1 Year. Analyzed by infused dose, above or below the median. The GMFM-66 is a clinical tool used to evaluate gross motor function in children with cerebral palsy and is scored using a propriety software program called the Gross Motor Ability Estimator (GMAE) that produces an interval level continuous score ranging from 0 to 100. Higher scores indicate better motor function. A negative change in GMFM-66 score indicates a reduction in motor function, a positive change indicates improvement in motor function, and zero indicates no change in motor function.
Time Frame: 1 Year
Population: Patients randomized to Autologous Umbilical Cord Blood were divided into two groups for this analysis: Low and High dose. The median dose infused in these 32 patients was used as the cut point to define Low and High doses: 1.98x10e7 total nucleated cells per kilogram of patient weight (TNCC/kg).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous UCB Reinfusion First, Then Placebo | Placebo First, Then Autologous UCB Reinfusion
Number analyzed (Participants) | 32 | 31
units on a scale
  All | 6.5 [-3 to 19] | 6.0 [-5 to 19]
  Low Infused Dose: number analyzed (Participants) | 16 | 0
  Low Infused Dose | 4 [-3 to 19] |
  High Infused Dose: number analyzed (Participants) | 16 | 0
  High Infused Dose | 8.5 [0 to 19] |
Statistical Analysis 1: Comparison: Autologous UCB Reinfusion First, Then Placebo; H0: The population distribution of the 1-year GMFM-66 change score is the same for patients infused with Low and High doses of autologous umbilical cord blood; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The population distribution of the 1-year GMFM-66 change score is the same for patients infused with High doses of autologous umbilical cord blood and Placebo; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Autologous UCB Reinfusion First, Then Placebo vs Placebo First, Then Autologous UCB Reinfusion; H0: The population distribution of the 1-year GMFM-66 change score is the same for patients infused with Low doses of autologous umbilical cord blood and placebo; Test type: Superiority; p = 0.21, Wilcoxon (Mann-Whitney)

28. Post Hoc Outcome: Observed Minus Expected GMFM-66 Change Score of All Subjects Receiving Autologous UCB and Who Are Greater Than or Equal to 2 Years of Age
Description: Validated functional curves were used to identify the expected 1-year change in GMFM-66 score given each child's age and Gross Motor Function Classification System (GMFCS) Level at baseline. The difference between observed change (in this study) and expected change was then calculated for each participant. The threshold defining Low/High dose is the median dose infused in all 63 enrolled patients, 2x10e7 TNCC/kg.
Time Frame: 1 year post-infusion with autologous umbilical cord blood
Population: Patients who received cord blood at baseline and 1 year post-infusion with Placebo, and who are >=2 years old (to allow calculation of expected GMFM-66 change scores from published data). An additional 6 are excluded because change scores were not observable due to subject withdrawal (5) or inability to comply due to a broken leg (1).
Measure: Median (Full Range); unit: units on a scale
Groups:
- Autologous Umbilical Cord Blood Reinfusion: Patients will be randomized to receive their autologous umbilical cord blood cells first or placebo first. Subjects will receive both infusions but will be randomized and blinded by which they are receiving first and second.
Arm/Group | Autologous Umbilical Cord Blood Reinfusion
Number analyzed (Participants) | 46
units on a scale
  All | 1.1 [-8.1 to 15.4]
  Low Infused Dose: number analyzed (Participants) | 23
  Low Infused Dose | -1.1 [-8.1 to 12.9]
  High Infused Dose: number analyzed (Participants) | 23
  High Infused Dose | 3.6 [-5.6 to 15.4]
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion; H0: The population distribution of differences between observed and expected GMFM-66 change scores at 1-year post-infusion is the same for patients receiving Low and High doses of autologous umbilical cord blood; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

29. Post Hoc Outcome: Peabody Gross Motor Quotient Change Score 1 Year After Receiving Autologous UCB.
Description: The Peabody Developmental Motor Scales - Second Edition (PDMS-2), Gross Motor Quotient change score was calculated for each patient at 1 year after infusion with autologous umbilical cord blood. Analyzed by infused dose, above or below the median. The Gross Motor Quotient score from the PDMS-2 was used in this study to evaluate gross motor function. The Gross Motor Quotient measures the ability to use large muscle systems for locomotion, maintain a stable posture when not moving, and throw/catch objects. The range of possible scores is 41 to 164. High scores indicate better gross motor function. Lower scores indicate less gross motor function ability.
Time Frame: 1 year post-infusion with autologous umbilical cord blood
Population: This group combines patients who received Autologous Umbilical Cord Blood at baseline or 1 year post-infusion with Placebo, and who are within the age range specified for the PDMS-2. The threshold defining Low/High dose is the median dose infused in all 63 enrolled patients, 2x10e7 TNCC/kg.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Autologous Umbilical Cord Blood Reinfusion
Number analyzed (Participants) | 47
units on a scale
  Low Infused Dose: number analyzed (Participants) | 25
  Low Infused Dose | 0 [-10 to 15]
  High Infused Dose: number analyzed (Participants) | 22
  High Infused Dose | 3 [-8 to 20]
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion; Test type: Superiority — H0: The population distribution of the Peabody Gross Motor Quotient change score 1 year post-infusion with autologous umbilical cord blood is the same in patients receiving a Low infused dose and a High infused dose; p = 0.03, Wilcoxon (Mann-Whitney)

30. Post Hoc Outcome: Change in Whole Brain Connectivity Measured by Diffusion Tensor Magnetic Resonance Imaging (MRI) of All Subjects 1 Year Post-infusion With Autologous UCB
Description: Change in whole brain connectivity measured by diffusion tensor magnetic resonance imaging (MRI). Changes in connectivity are normalized to white matter volume.
Time Frame: 1 year post-infusion with autologous umbilical cord blood
Population: This group combines patients who received Autologous Umbilical Cord Blood whether at baseline or 1 year post-infusion with Placebo and is limited to patients without morphologic brain abnormalities that prevented accurate anatomical image parcellation. Low/High dose is defined as the median dose infused in all 63 enrolled patients, 2x10e7 TNCC/kg.
Measure: Mean (Standard Deviation); unit: Number of connections x10e5
Groups:
- Autologous Umbilical Cord Blood Reinfusion: All participants will be treated with autologous cord blood reinfusion, but the time course will vary between groups and participants will be blinded to the order in which they receive infusions.
  Autologous Umbilical Cord Blood or Placebo: All participants will be treated with autologous cord blood reinfusion, but the time course will vary between groups and participants will be blinded to the order in which they receive infusions. Patients will be randomized to receive their autologous umbilical cord blood cells first or placebo first. Subjects will receive both infusions but will be randomized and blinded by which they are receiving first and second.
Arm/Group | Autologous Umbilical Cord Blood Reinfusion
Number analyzed (Participants) | 38
Number of connections x10e5
  Low Infused Dose: number analyzed (Participants) | 19
  Low Infused Dose | 0.10 (0.32)
  High Infused Dose: number analyzed (Participants) | 19
  High Infused Dose | 0.30 (0.24)
Statistical Analysis 1: Comparison: Autologous Umbilical Cord Blood Reinfusion; H0: The true mean 1-year change in normalized whole brain connectivity is the same in patients infused with Low and High doses of autologous umbilical cord blood; Test type: Superiority; p = 0.04, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.01 to 0.38]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Since there is no washout period for autologous umbilical cord blood transfusions, the only adverse events included in the placebo arm were those events that occurred in subjects that had not yet received cord blood. All other adverse events that occurred in subjects that had been exposed to cord blood at either Baseline or Year 1 were included in the "Autologous Umbilical Cord Blood" arm.
Groups:
- Placebo: All participants will be treated with autologous cord blood reinfusion, but the time course will vary between groups and participants will be blinded to the order in which they receive infusions.
  Autologous Umbilical Cord Blood or Placebo: All participants will be treated with autologous cord blood reinfusion, but the time course will vary between groups and participants will be blinded to the order in which they receive infusions. Patients will be randomized to receive their autologous umbilical cord blood cells first or placebo first. Subjects will receive both infusions but will be randomized and blinded by which they are receiving first and second.
Arm/Group | Autologous Umbilical Cord Blood Reinfusion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/63
Other Adverse Events (participants affected / at risk) | 24/63 | 4/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Umbilical Cord Blood Reinfusion (N=63) | Placebo (N=63)
Flushed in face with hypersensitivity rash on trunk (Endocrine disorders) | 0 (0) | 1 (1) — Subject developed polydipsia, polyuria, and hyperglycemia the evening after infusion and was seen in the ED. Subject was diagnosed with type I diabetes (mother also has type I diabetes). This was reported to Medwatch.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Umbilical Cord Blood Reinfusion (N=63) | Placebo (N=63)
Flushed in face with hypersensitivity rash on trunk. Sats 92%. No wheezing. Benadryl given (Immune system disorders) | 0 (0) | 1
Tactile temp overnight. Left otitis media (Infections and infestations) | 0 (0) | 1
Painful urination and spotting 1 wk post infusion. (Renal and urinary disorders) | 1 | 0 (0) — Seen by urgent care-abx started, stopped when cultures neg.
Admitted to ER with polyuria and polydipsia (Metabolism and nutrition disorders) | 1 | 0 (0) — Highest blood sugar 757. Received fluid and insulin- Diabetes Dx
Rash on abdomen and legs. No itching or welps. No treatment- resolved next day (Skin and subcutaneous tissue disorders) | 0 (0) | 1
Fever of 102 3 days post. Negative culture. No treatment-resolved in 3 days. (General disorders) | 1 | 0 (0)
Stomach pain from hydronephrotic dysplastic kidney (Gastrointestinal disorders) | 1 | 0 (0)
G tube fell out (Gastrointestinal disorders) | 1 | 0 (0)
Pneumonia-hospitalized 10 days (Infections and infestations) | 1 | 0 (0)
Flu (Infections and infestations) | 1 | 0 (0)
Fractured left foot (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
Withdrawn during strep throat and sinus infection- EEG showed spikes , but no epileptiform activity (Infections and infestations) | 1 | 0 (0)
Febrile seizure-isolated, not treated (Nervous system disorders) | 1 | 0 (0)
G tube placement (Gastrointestinal disorders) | 0 (0) | 1
Fever 2 weeks post infusion-found to be viral laryngitis (Infections and infestations) | 1 | 0 (0)
Admitted to hospital- Flu (Infections and infestations) | 1 | 0 (0)
Cough/Cold requiring antibiotics (Infections and infestations) | 1 | 0 (0)
Pneumonia requiring antibiotics (Infections and infestations) | 1 | 0 (0)
Developed cough and sats fell to 70 toward end of MRI- received blow by O2 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Adverse behavioral rxn to Benadryl given infusion day- crying (General disorders) | 1 | 0 (0)
Diagnosed with Cockayne syndrome (Congenital, familial and genetic disorders) | 1 | 0 (0)
Ear infection, cough, and fever 2 wks post infusion (Infections and infestations) | 1 | 0 (0)
Fever for 2 days prior to infusion-given Tylenol (General disorders) | 1 | 0 (0)
Right foot fracture- cast required (Musculoskeletal and connective tissue disorders) | 1 | 0 (0)
High fever and febrile seizure associated with viral infection at home 2 weeks post infusion (Nervous system disorders) | 1 | 0 (0)
Febrile Seizure (Nervous system disorders) | 1 | 0 (0)
2 seizures in interval- due to virus- on anti-seizure med (Nervous system disorders) | 1 | 0 (0)
Briefly hospitalized for bronchiolitis and dehydration- treated with rocephin and rehydration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Ear infection (Infections and infestations) | 1 | 0 (0)
Agitation and mild conjunctivitis of right eye following infusion. (Immune system disorders) | 1 | 0 (0) — Returned to baseline after being given Benadryl.
Inhaler needed for respiratory wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 (0)
Diagnosed with walking pneumonia prior to final visit- on antibiotics (Infections and infestations) | 0 (0) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No